CLINICAL TRIAL: NCT04604561
Title: Physician Initiated Evaluation of EnVisio SmartClip for Intraoperative Localization of Breast Masses
Brief Title: Evaluation of EnVisio SmartClip for Intraoperative Localization of Breast Masses
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Elucent Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-20335
Record Dates: First submitted 2020-10-09; First posted 2020-10-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: SmartClip; EnVisio™ Navigation System
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Participants receiving SmartClip: Participants will undergo a preoperative physical exam and at least one preoperative ultrasound demonstrating the mass for resection. The SmartClip will be placed under ultrasound guidance. Post-placement mammogram will be obtained after placement of the clip. The SmartClip can be placed up to 30 days prior to the planned surgical resection. At the time of definitive surgery, the Envisio system will be used to identify the clip and the targeted lesion for resection. Intraoperatively, a specimen radiograph will be performed to confirm the presence of the SmartClip and the targeted lesion in the surgical specimen. The breast surgical specimen will be sent for gross examination, including measurements of the tumor in 3 axes. Immediately post-procedure, the performing surgeon will fill out a questionnaire to determine the ability of localizing in-breast lesions using the Envisio Navigation and SmartClip system in surgery.
  Interventions: Device: EnVisio SmartClip; Device: EnVisio™ Navigation System
- Radiologist Placing SmartClip: Radiologist will place SmartClip under ultrasound guidance. A Post-placement mammogram will be obtained after placement of the SmartClip. Immediately post-procedure, the performing radiologist will fill out a questionnaire.
  Interventions: Device: EnVisio SmartClip; Device: EnVisio™ Navigation System
- Surgeon: The surgeon will use the EnVisio™ Navigation System to identify the SmartClip and the targeted lesion for resection. Immediately post-procedure, the performing surgeon will fill out a questionnaire
  Interventions: Device: EnVisio SmartClip; Device: EnVisio™ Navigation System

INTERVENTIONS:
Device: EnVisio SmartClip — The Envisio SmartClip is an FDA-cleared (approved) device for localization of in-breast lesions. While using The EnVisio™ Navigation System, the system will detect the presence of the SmartClip™ Soft Tissue Marker(s) and provide real-time three-dimensional navigation during the surgery.
Device: EnVisio™ Navigation System — The EnVisio™ Navigation System acquires and analyzes electromagnetic signatures that display the relative distance, depth, and direction from the tip of the electrosurgical tool to the implanted SmartClipTM(s) within the surgeon's field of view during the procedure.

SUMMARY:
This is a pilot study to estimate the success of the SmartClip device for accurate placement and reproducibility of intraoperative identification of in-breast lesions and for excision utilizing surgical navigation indicators.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least one and up to 3 sonographically or mammographically identifiable in-breast or axillary targets and consent to undergo a surgical resection using the SmartClip localization system at the McKinley operative suites at Moffitt Cancer Center. Multiple sites for localization may be used, up to a maximum of 3 SmartClips per patient. Mammographically or sonographically visible biopsy clips may be used as a localizing target.
* Participants must be age > or = 18 years.

Exclusion Criteria:

* Participants with sonographically or mammographically occult target lesions
* Participants with greater than 35cm chest to bust depth
* Participants undergoing mastectomy for resection of the targeted lesion
* Inability to undergo surgery at the McKinley OR suites due to institutional anesthesia guidelines
* Patients requiring use of more than 3 SmartClips to localize targets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited to this study from the Moffitt Cancer Center Comprehensive Breast Clinic. Patients are seen in this clinic by breast surgeons from the Comprehensive Breast Program at Moffitt Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Ability of localizing in-breast lesions using the Envisio Navigation and SmartClip system in surgery - Radiologist Cohort | 1 year
  Questions 1,2,5,6,7 & 8 from the Radiologist survey will evaluate the EnVisio system for reproducible in-breast tumor localization by the performing physicians.
Ability of localizing in-breast lesions using the Envisio Navigation and SmartClip system in surgery - Surgeon Cohort | 1 year
  Questions 4, 5, 6, 8, 9, 10, & 11 from the Surgeon survey will evaluate the EnVisio system for reproducible in-breast tumor localization by the performing physicians.

SECONDARY OUTCOMES:
Placement of the SmartClip on preoperative imaging to clip location on specimen radiography | 1 year
  Radiologists will take radiologist questionnaire evaluating their experience using the SmartClip
Placement and visibility of the clip by breast radiologists | 1 year
  Radiologists will take radiologist questionnaire evaluating their experience using the SmartClip
Intraoperative use of the device system by surgeons | 1 year
  Surgeons will take surgeon questionnaire evaluating their experience using the SmartClip and EnVisio™ Navigation System
Surgical outcomes with use of the SmartClip | 1 year
  Surgeons will take surgeon questionnaire evaluating their experience using the SmartClip and EnVisio™ Navigation System

CONTACTS AND LOCATIONS:
Overall Officials: M. Catherine Lee, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/